CLINICAL TRIAL: NCT01478958
Title: The Effects of the Substitution of Dietary SFA With n-6 PUFA or MUFA on Vascular Function
Brief Title: Dietary Intervention and Vascular Function
Acronym: DIVAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Julie Lovegrove, Professor, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: N02044
Record Dates: First submitted 2011-11-16; First posted 2011-11-23 (Estimated); Results first posted 2014-07-15 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-06

CONDITIONS: Cardiovascular Disease
Keywords: fatty acids; cardiovascular disease; vascular function; microparticles
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- high saturated fat diet (Active Comparator)
  Interventions: Dietary Supplement: SFA diet
- high monounsaturated fat diet (Experimental)
  Interventions: Dietary Supplement: MUFA diet
- high n-6 polyunsaturated fat diet (Experimental)
  Interventions: Dietary Supplement: n-6 PUFA diet

INTERVENTIONS:
Dietary Supplement: SFA diet — Volunteers are following a high saturated fat diet for a 4-month period
  Arms: high saturated fat diet
Dietary Supplement: MUFA diet — Volunteers are following a high monounsaturated fat diet for a 4-month period
  Arms: high monounsaturated fat diet
Dietary Supplement: n-6 PUFA diet — Volunteers are following a high n-6 polyunsaturated fat diet for a 4-month period
  Arms: high n-6 polyunsaturated fat diet

SUMMARY:
It is well established that diet plays an important role in both the development and progression of heart disease. Different types of dietary fat have varying effects on heart disease risk factors. The elasticity of an individual's blood vessels is strongly associated with heart disease risk and recent evidence suggests that dietary manipulation may influence elasticity of the blood vessels with dietary fat (including saturated, monounsaturated and polyunsaturated fatty acids) as a potentially important modulator. Substantial evidence exists on the effects of monounsaturated fats (type of fatty acids mainly found in olive and rapeseed oil), n-6 polyunsaturated fats (type of polyunsaturated fatty acids found in vegetable oils) and saturated fat (found mainly in animal derived products) on lipid levels. However, the influence of these dietary fats on the elasticity of blood vessels remains unclear.The main purpose of the DIVAS study is to determine the effects of the substitution of saturated fats with either n-6 polyunsaturated or monounsaturated fats on blood vessel elasticity and to determine the effects of these different dietary fats on other risk factors for heart disease including lipoproteins and inflammatory biomarkers.

ELIGIBILITY:
Inclusion Criteria:

Adults should have a relative risk (RR) of > 1.5 of developing cardiovascular disease (CVD) based on presenting with at least one recognised risk factor for CVD:

* total cholesterol (TC) > 6.0 mmol/l
* HDL cholesterol (HDLC) ≤ 1.0 mmol/l male, ≤ 1.3 mmol/l female
* Glucose ≥ 6 mmol/l
* Stage 1 hypertension or above i.e. a systolic BP ≥ 140 mmHg, diastolic BP ≥ 90 mmHg
* BMI 28-35 kg/m2
* waist >102 cm male or > 84 cm female
* Adults with a first degree relative with either a history of premature CVD - age of onset younger than 55 y in fathers, sons or brothers or younger than 65 y in mothers, daughters or sisters, or type 2 diabetes.

Exclusion Criteria:

* having suffered a myocardial infarction/stroke in the past 12 months
* diabetic (diagnosed or fasting glucose > 7 mmol/l) or suffer from other endocrine disorders
* suffering from renal or bowel disease or have a history of choleostatic liver or pancreatitis
* on drug treatment for hyperlipidaemia, hypertension, inflammation or hypercoagulation
* no history of alcohol abuse
* planning or on a weight reducing regime
* taking any fish oil, fatty acid or vitamin and mineral supplements
* pregnant, lactating or planning a pregnancy
* smokers

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 202 (Actual)
Dates: Start 2010-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Lovegrove, BSc PhD RNutr, Principal Investigator — University of Reading
Locations (2):
- United Kingdom (2):
  - Department of Food and Nutritional Sciences, University of Reading, Reading, Berkshire
  - University of Reading, Reading, Berkshire

REFERENCES:
- [Derived] Sellem L, Eichelmann F, Jackson KG, Wittenbecher C, Schulze MB, Lovegrove JA. Replacement of dietary saturated with unsaturated fatty acids is associated with beneficial effects on lipidome metabolites: a secondary analysis of a randomized trial. Am J Clin Nutr. 2023 Jun;117(6):1248-1261. doi: 10.1016/j.ajcnut.2023.03.024. Epub 2023 Apr 11. PMID 37062359
- [Derived] Weech M, Altowaijri H, Mayneris-Perxachs J, Vafeiadou K, Madden J, Todd S, Jackson KG, Lovegrove JA, Yaqoob P. Replacement of dietary saturated fat with unsaturated fats increases numbers of circulating endothelial progenitor cells and decreases numbers of microparticles: findings from the randomized, controlled Dietary Intervention and VAScular function (DIVAS) study. Am J Clin Nutr. 2018 Jun 1;107(6):876-882. doi: 10.1093/ajcn/nqy018. PMID 29741564
- [Derived] Shatwan IM, Weech M, Jackson KG, Lovegrove JA, Vimaleswaran KS. Apolipoprotein E gene polymorphism modifies fasting total cholesterol concentrations in response to replacement of dietary saturated with monounsaturated fatty acids in adults at moderate cardiovascular disease risk. Lipids Health Dis. 2017 Nov 23;16(1):222. doi: 10.1186/s12944-017-0606-3. PMID 29169396
- [Derived] Vafeiadou K, Weech M, Altowaijri H, Todd S, Yaqoob P, Jackson KG, Lovegrove JA. Replacement of saturated with unsaturated fats had no impact on vascular function but beneficial effects on lipid biomarkers, E-selectin, and blood pressure: results from the randomized, controlled Dietary Intervention and VAScular function (DIVAS) study. Am J Clin Nutr. 2015 Jul;102(1):40-8. doi: 10.3945/ajcn.114.097089. Epub 2015 May 27. PMID 26016869
- [Derived] Weech M, Vafeiadou K, Hasaj M, Todd S, Yaqoob P, Jackson KG, Lovegrove JA. Development of a food-exchange model to replace saturated fat with MUFAs and n-6 PUFAs in adults at moderate cardiovascular risk. J Nutr. 2014 Jun;144(6):846-55. doi: 10.3945/jn.114.190645. Epub 2014 Apr 9. PMID 24717370

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited in three cohorts between November 2009 and June 2012.
Groups:
- High Saturated Fat Diet: SFA diet: Volunteers followed a high saturated fat diet for a 4-month period
- High Monounsaturated Fat Diet: MUFA diet: Volunteers followed a high monounsaturated fat diet for a 4-month period
- High n-6 Polyunsaturated Fat Diet: n-6 PUFA diet: Volunteers followed a high n-6 polyunsaturated fat diet for a 4-month period
Period: Overall Study
Arm/Group | High Saturated Fat Diet | High Monounsaturated Fat Diet | High n-6 Polyunsaturated Fat Diet
Started | 67 | 66 | 69
Completed | 65 | 64 | 66
Not Completed | 2 | 2 | 3
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Weight loss | 1 | 0 | 0
Not completed — Re-located | 0 | 1 | 0
Not completed — Unable to comply | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Saturated Fat Diet | High Monounsaturated Fat Diet | High n-6 Polyunsaturated Fat Diet | Total
Number analyzed (Participants) | 65 | 64 | 66 | 195
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (9) | 43 (11) | 45 (10) | 44 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 37 | 37 | 110
  Male | 29 | 27 | 29 | 85
Region of Enrollment [Number; unit: participants]
  United Kingdom | 65 | 64 | 66 | 195
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.7 (4.4) | 26.3 (3.9) | 27.0 (3.7) | 26.7 (4.0)
Waist Circumference [Mean (Standard Deviation); unit: cm] | 92.1 (12.1) | 88.2 (10.3) | 92.1 (13.1) | 90.9 (12.0)
24-hour Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mm Hg] | 121 (12) | 121 (10) | 124 (11) | 122 (11)
24-hour Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mm Hg] | 75 (8) | 74 (6) | 76 (8) | 75 (7)
Fasting Total Cholesterol (TC) [Mean (Standard Deviation); unit: mmol/L] | 5.38 (0.98) | 5.43 (1.07) | 5.57 (1.27) | 5.46 (1.09)
Fasting High-Density Lipoprotein Cholesterol (HDL-C) [Mean (Standard Deviation); unit: mmol/L] | 1.45 (0.33) | 1.48 (0.39) | 1.51 (0.38) | 1.48 (0.37)
Ratio of TC:HDL-C [Mean (Standard Deviation)] | 3.92 (1.20) | 3.85 (0.99) | 3.85 (1.12) | 3.87 (1.10)
Fasting Low-Density Lipoprotein Cholesterol (LDL-C) [Mean (Standard Deviation); unit: mmol/L] | 3.67 (0.93) | 3.71 (0.88) | 3.81 (1.13) | 3.73 (0.98)
Fasting Triacylglycerol (TAG) [Mean (Standard Deviation); unit: mmol/L] | 1.31 (0.77) | 1.18 (0.53) | 1.26 (0.67) | 1.25 (0.67)
Fasting Glucose [Mean (Standard Deviation); unit: mmol/L] | 5.09 (0.43) | 5.00 (0.45) | 5.05 (0.44) | 5.05 (0.44)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Flow Mediated Dilatation (FMD)
Time Frame: Baseline, 4 months
Population: Number of participants analyzed: n=171. n=24 were images of poor quality that could not be analyzed successfully.
Measure: Mean (Standard Error); unit: post-occlusion diameter change as %
Arm/Group | High Saturated Fat Diet | High Monounsaturated Fat Diet | High n-6 Polyunsaturated Fat Diet
Number analyzed (Participants) | 59 | 57 | 55
post-occlusion diameter change as % | -0.39 (0.24) | -0.07 (0.32) | -0.08 (0.31)
Statistical Analysis 1: Comparison: High Saturated Fat Diet vs High Monounsaturated Fat Diet vs High n-6 Polyunsaturated Fat Diet; To detect a 2% inter-group difference in FMD (primary outcome) using a SD of 2.3, 90% power and 5% significance level, n=171 participants were required (n=57 per group), increasing to n=228 to include a 25% dropout rate; Test type: Superiority or Other; p = 0.238, General Linear Model Univariate Analysis — Overall diet effect. No post-hoc analyses required. Adjusted for multiple comparisons; Baseline values for %FMD, BMI, age, gender and intervention diet used as prognostic factors in model
Statistical Analysis 2: Comparison: High Saturated Fat Diet; Test type: Superiority or Other; p = 0.021, General Linear Model Univariate Analysis — Effect of the SFA-rich diet relative to baseline; Baseline values for %FMD, BMI and age, gender and intervention diet were used as prognostic factors in the model
Statistical Analysis 3: Comparison: High Monounsaturated Fat Diet; Test type: Superiority or Other; p > 0.05, General Linear Model Univariate Analysis — Effect of MUFA-rich diet relative to baseline; Baseline values for %FMD, BMI and age, gender and intervention diet were used as prognostic factors in the model
Statistical Analysis 4: Comparison: High n-6 Polyunsaturated Fat Diet; Test type: Superiority or Other; p > 0.05, General Linear Model Univariate Analysis — Effect of n-6 PUFA-rich diet relative to baseline; Baseline values for %FMD, BMI and age, gender and intervention diet were used as prognostic factors in the model

2. Secondary Outcome: Cardiovascular Risk Factors (Lipids, Inflammatory Markers, Indices of Insulin Resistance, Cell Microparticles, Endothelial Progenitor Cells)
Description: Data for fasting serum lipids (total cholesterol (TC), high-density lipoprotein cholesterol (HDL-C), TC:HDL-C ratio, low-density lipoprotein cholesterol (LDL-C), triacylglycerol (TAG)).
Time Frame: 4 months
Reporting Status: Not Posted

3. Secondary Outcome: 24-hour Ambulatory Blood Pressure
Description: 24-hour, daytime and night-time measures of systolic blood pressure (SBP), diastolic blood pressure (DBP), pulse pressure (PP; SBP-DBP) and heart rate (HR)
Time Frame: 4 months
Reporting Status: Not Posted

4. Secondary Outcome: Vascular Stiffness by Pulse Wave Velocity (PWV), Pulse Wave Analysis (PWA) and Digital Volume Pulse (DVP)
Description: PWV (m/s) PWA produces Augmentation Index (AIx; %) DVP produces Stiffness Index (SI; m/s) and Reflection Index (RI; %)
Time Frame: 4 months
Reporting Status: Not Posted

5. Secondary Outcome: Microvascular Reactivity (Laser Doppler Imaging With Iontophoresis)
Description: Laser Doppler imaging (LDI) with iontophoresis of acetylcholine (Ach; endothelium-dependent vasodilation) and sodium nitroprusside (SNP; endothelium-independent vasodilation).
Time Frame: 4 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | High Saturated Fat Diet | High Monounsaturated Fat Diet | High n-6 Polyunsaturated Fat Diet
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/66 | 0/69
Other Adverse Events (participants affected / at risk) | 0/67 | 0/66 | 0/69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No